CLINICAL TRIAL: NCT03560219
Title: AssociatioN of Genetic Polymorphisms With ATrial fibrOsis and Thrombogenic Substrate in Patients With Non-vaLvular atrIAl Fibrillation
Acronym: ANATOLI-AF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Memorial Ankara Hospital (Other)
Responsible Party: Principal Investigator, Sercan Okutucu, Associate Professor, Memorial Ankara Hospital
Other Study IDs: MANK200801
Record Dates: First submitted 2018-06-06; First posted 2018-06-18 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Atrial Fibrillation; Thrombosis; Stroke; Genetic Predisposition; Heart Diseases
Keywords: Atrial Fibrillation; Atrial Fibrosis; Genome Wide Association Studies; Biomarkers; Echocardiography; Magnetic Resonance Imaging; Flow Mediated Dilatation; Thrombogenic Substrate
MeSH Terms: conditions — Atrial Fibrillation; Thrombosis; Stroke; Genetic Predisposition to Disease; Heart Diseases | interventions — Echocardiography; Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Biomarkers, Cardiac Magnetic Resonance Imaging, Echocardiography, Flow Mediated Dilatation, Genetic Analysis — Key variables that will be recorded include the following:
  * Clinical
    * Age
    * Gender
    * BMI
    * Diabetes Mellitus
    * Hypertension
    * Heart Failure
    * Ischemic Stroke / TIA
    * Thromboembolism
    * Coronary Artery Disease
    * Peripheral Arterial Disease
    * Glomerular Filtration Rate
  * Contrast-enhanced MRI
    o Presence and extent of atrial fibrosis
  * Biomarkers
    * IL-6
    * CRP
    * D-dimer
    * Fibrinogen
  * Transthoracic Echocardiography
    * LA Volume Index (LAVI)
    * LA Strain, Global
    * LA Strain rate, Positive peak, Global
    * LA Strain rate, early negative peak, Global
    * LA Strain rate, late negative peak, Global
    * LA Emptying Fraction (LAEF)
    * LVH
    * LVEF
  * Endothelial function o FMD

SUMMARY:
Atrial fibrillation (AF) is the most frequently encountered cardiac arrhythmia. Emerging data suggests that common genetic variants are associated with the development of AF. The main feature of the structural remodelling in AF is atrial fibrosis and is considered the substrate for AF perpetuation. Genome-wide association studies suggest that AF-susceptibility variants may modulate atrial fibrosis. However, the association between atrial fibrosis and genetic polymorphisms in humans has not yet been specifically investigated. In this study, we plan to investigate the relationship between genetic polymorphisms, atrial fibrosis and other components of thrombogenic substrate in patients with non-valvular AF. Primary objectives of this study are to assess associations between (i) polymorphic genetic variants and atrial fibrosis (detected by magnetic resonance imaging), (ii) polymorphic genetic variants and components of thrombogenic substrate (inflammation, endothelial function, prothrombotic state, atrial functions).

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most frequently encountered cardiac arrhythmia. Emerging data suggests that common genetic variants are associated with the development of AF. The main feature of the structural remodelling in AF is atrial fibrosis and is considered the substrate for AF perpetuation. Genome-wide association studies suggest that AF-susceptibility variants may modulate atrial fibrosis. However, the association between atrial fibrosis and genetic polymorphisms in humans has not yet been specifically investigated. In this study, we plan to investigate the relationship between genetic polymorphisms, atrial fibrosis and other components of thrombogenic substrate in patients with non-valvular AF. Primary objectives of this study are to assess associations between (i) polymorphic genetic variants and atrial fibrosis (detected by magnetic resonance imaging), (ii) polymorphic genetic variants and components of thrombogenic substrate (inflammation, endothelial function, prothrombotic state, atrial functions). Patients are planned to be recruited from four major cardiology departments: Memorial Ankara Hospital, Ministry of Health Subspecialty Training Hospital of Turkey, Ufuk University and Gazi University hospitals. Key variables that will be recorded include the clinical, contrast-enhanced MRI, biomarkers, echocardiographic and assessment of endothelial function. All statistical analyses will be conducted using Stata version 11.0 (StataCorp, College Station, TX). Univariate and multivariate regression models will be used to determine the odds ratio of each variable to assess the association of the clinical and laboratory parameters, and genotype profiles with the presence of LA fibrosis. Furthermore, data mining methods like support vector machines and/or random forests are planned to be used for detecting the impact of each potential predictor on the risk of LA fibrosis. Additionally, to determine the effect of different alleles of the identified risk SNPs, 2-way and 3-way multi dimensionality reduction (MDR) analysis will be performed. Bioinformatics investigations to determine SNP-SNP, SNP-gene and SNP-Phenotype interactions will be performed by combined p-value and biological network analysis.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Documented AF
* Paroxysmal and persistent AF

Exclusion Criteria:

* Patients with infectious or non-infectious inflammatory disease
* Patients with structural heart disease
* Acute coronary syndrome
* Severe liver and kidney dysfunction
* Cancer
* Immune disorders
* Surgery and stroke within six months

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population will include patients with documented AF (Paroxysmal or Persistent) over the age of 18. Patients are planned to be recruited from four major cardiology departments: Memorial Ankara Hospital, Ministry of Health Subspecialty Training Hospital of Turkey, Ufuk University and Gazi University hospitals.
Sampling Method: Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Associations between polymorphic genetic variants and atrial fibrosis | Through study completion, an average of 1 year
  (detected by MRI)
Associations between polymorphic genetic variants and components of thrombogenic substrate | Through study completion, an average of 1 year
  Thrombogenic substrate (inflammation, endothelial function, prothrombotic state, atrial functions)

IPD SHARING:
Plan to Share IPD: No